CLINICAL TRIAL: NCT00866879
Title: Randomized Conversion of Calcineurin-Inhibitors(Tacrolimus to Sirolimus),6-24 Months Post Transplant Prednisone-Free Immunosuppression Regimen: Impact of Incidence of Acute Cellular Rejection,Renal Allograft Function & Lymphocytes Function
Brief Title: Randomized Conversion of Calcineurin-Inhibitors in Renal Allograft Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Lorenzo Gallon, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU8308 0773-017; 0468H1-4472 (Other: Pfizer (Wyeth))
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Renal Transplant Rejection
Keywords: Sirolimus; Rapamune; Immunosuppression; Renal allograft function; Lymphocytes function
MeSH Terms: interventions — Sirolimus; Demography; Health Records, Personal; Blood Specimen Collection; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Group 1 will continue immunosuppression medication per standard of care (SOC) at Northwestern by taking mycophenolate mofetil and tacrolimus.
  Interventions: Other: Demographic Data, Medical History, and Donor Data; Procedure: Blood Draws for Control Group; Procedure: Kidney Biopsy
- Transition to Sirolimus Group (Experimental): Group 2 will switch immunosuppression medication to taking mycophenolate mofetil and sirolimus
  Interventions: Drug: Sirolimus; Other: Demographic Data, Medical History, and Donor Data; Procedure: Blood Draws for Experimental Group; Procedure: Kidney Biopsy
- Donors (Other): Data and blood samples from the donors are collected in this study to contribute to the general knowledge to be used in assessing the two donor recipient groups, which are the target of this study.
  Interventions: Procedure: Donor Blood Draws; Other: Donor Information

INTERVENTIONS:
Drug: Sirolimus — Sirolimus will initially be given at a dose of 2-4 mg orally (PO) daily. The dose will be modified to achieve 24 hours trough concentrations of 6-10 ng/ml by high-performance liquid chromatography (HPLC) assay. This medication will be given in an open label fashion. The first dose of sirolimus will be given at the time of randomization to those patients assigned to have tacrolimus switched to sirolimus.
  Other Names: Rapamune
  Arms: Transition to Sirolimus Group
Other: Demographic Data, Medical History, and Donor Data — Age at transplant, sex, race, cause of end-stage renal disease, medical history, donor age, cadaveric vs. living kidney transplant, histocompatibility/cross match data, viral serology, history of acute rejection and delayed graft function, use of induction therapy and immunosuppressants, use of Angiotensin Converting Enzyme Inhibitor (ACEI) and/or Angiotensin Receptor Blockers (ARB) level of renal allograft function-estimated GFR (e-GFR(12) using Modification of Diet in Renal Disease (MDRD) formula, proteinuria.
  Arms: Control; Transition to Sirolimus Group
Procedure: Blood Draws for Control Group — Subjects maintaining standard of care drug treatment of TAC and MMF will have monthly labs in addition to the baseline pre-randomization labs, at 6, 12, and 24 Months post-randomization. Peripheral blood leukocytes will be obtained.
  Arms: Control
Procedure: Blood Draws for Experimental Group — This group will have monthly labs taken but will also have weekly labs during the period of conversion to monitor renal function and bone marrow function. In addition to the baseline pre-randomization labs, and labs collected at 6, 12, and 24 Months post-randomization, peripheral blood leukocytes will be obtained.
  Arms: Transition to Sirolimus Group
Procedure: Donor Blood Draws — Peripheral blood leukocytes from living donors obtained at the time of randomization. These donor leukocytes will be used as stimulator cells to study the functional activity of the recipient's lymphocytes function.
  Arms: Donors
Other: Donor Information — Donor age, cadaveric vs. living donor, and histocompatibility and cross match to recipient
  Arms: Donors
Procedure: Kidney Biopsy — Kidney biopsy at 24 Months to compare to the standard of care biopsy taken at 12 Months. This information will help evaluate renal allograft pathology and renal allograft tissue gene expression profiles of the two groups. Renal allograft biopsies will be stored in RNA later (preservative) to further extend knowledge on the effect of calcineurin-inhibitors (CI) free immunosuppression on gene expression profiles.
  Arms: Control; Transition to Sirolimus Group

SUMMARY:
This study is being done to investigate the impact of changing immunosuppressive medications from tacrolimus (Prograf®) to sirolimus (Rapamune®) between 6 and 24 months post transplant. The primary purpose of this research study is to evaluate whether the use of mycophenolate mofetil(MMF)/Cellcept® and tacrolimus(TAC)/Prograf® (Group 1) or mycophenolate mofetil(MMF)/Cellcept® and sirolimus/Rapamune® (Group 2) impacts the incidence of acute cellular rejection in post kidney transplant patients. This study will examine whether switching from tacrolimus to sirolimus will better preserve long-term kidney function.

DETAILED DESCRIPTION:
For this research study, between 6 and 24 Months post-transplant, we plan to prospectively randomize 2:1 renal transplant patients to either:

* Substitute tacrolimus (TAC) with sirolimus and continue mycophenolate mofetil (MMF) or
* Continue with tacrolimus (TAC) and mycophenolate mofetil (MMF)

A total of 400 patients are expected to be screened for the randomization. We expect to randomize 275 renal transplant patients into this protocol (275 donors to be recruited).

The following data will be collected at the time of randomization:

Recipient demographics: (i) age at transplantation, (ii) sex, and (iii) race.

Clinical history: (i) causes of end-stage renal disease, and (ii) past medical history.

Transplant related information: (i) donor age, (ii) cadaveric versus living kidney transplant, (iii) histocompatibility and cross match data, (iv) viral serology, (v) history of acute rejection and delayed graft function, (vi) use of induction therapy and immunosuppressants, (vii) use of ACEI and/or ARB, and (viii) level of renal allograft function-estimated GFR (e-GFR(12) using MDRD formula, proteinuria.

Peripheral blood leukocytes will be obtained from renal transplant recipients for baseline (prior to randomization) lymphocytes functional activity and characterization of lymphocytes subpopulations by flow cytometry analysis.

Peripheral donor leukocytes (from living donor patients) will also be obtained at the time of randomization. These donor leukocytes will be used as stimulator cells to study the functional activity of the recipient's lymphocytes function.

The recipients assigned to continue with tacrolimus and MMF will be routinely followed at the outpatient Comprehensive Transplant Center (CTC) with monthly labs. In addition to labs at baseline pre-randomization, 6, 12 and 24 Months post-randomization, peripheral blood leukocytes will be obtained to study lymphocytes functional activity and to characterize lymphocytes subpopulations by flow cytometry analysis.

Post randomization: The recipients assigned to switch from tacrolimus to sirolimus and continue with MMF will be routinely followed at the CTC with monthly labs. During the period of conversion from tacrolimus to sirolimus, weekly labs will be obtained to monitor renal function and bone marrow function. In addition to labs at baseline pre-randomization, 6, 12 and 24 Months post-randomization, peripheral blood leukocytes will be obtained to study lymphocytes functional activity to characterize lymphocytes subpopulations by flow cytometry analysis. Urine will be collected to assess tubular toxicity by evaluating urinary biomarkers.

Both groups of patients will be followed for 2 years post-randomization. In addition to monitoring renal allograft function, we will evaluate the incidence of acute rejection, patient and graft survival, impact of CI conversion on the lipid profile, incidence of hypertension, malignancies, opportunistic infections, and post-transplant diabetes mellitus (DM). For those willing to undergo an optional kidney biopsy, one will be performed at the end of the second year in order to evaluate renal allograft pathology and renal allograft tissue gene expression profiles of the two groups.

With the peripheral leukocytes obtained at baseline prior to randomization and at 6, 12 and 24 Months post-randomization, we will investigate possible modifications of lymphocytes function and the lymphocytes subpopulations that might have occurred as a consequence of the switch from tacrolimus to sirolimus.

Obtaining renal allograft tissue samples at 24 months post randomization can have potential important ramifications to help explain the mechanisms of fibrosis and tubular atrophy typically associated with CI and the role of CI elimination with the substitution of sirolimus (SRL). All data will then be analyzed comparing gene expression profiles of peripheral blood (Pax gene tubes are routinely collected at the different time points as part of the original study). Based on power analysis, we will perform 24 months post randomization biopsies in 70% of the total subjects enrolled in the study (approximately 46 subjects from the tacrolimus/MMF group and approximately 93 subjects from the sirolimus/MMF group).

We plan to obtain renal allograft biopsies at 24 Months for those that consent for this additional biopsy. This will be compared to the standard of care 12 months post-transplant biopsy to allow us to address the effect of immunosuppressive modifications on renal allograft pathology at 24 months post randomization. Renal allograft biopsies will also be stored in RNA later to further extend our knowledge on the effect of CI free immunosuppression on gene expression profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should be adults ≥ 18- ≤ 70 years of age
2. Subjects can be either gender or of any ethnic background
3. Subjects should be single organ recipients (kidney only)
4. Subjects must be able to understand the protocol and provide informed consent.

Exclusion Criteria:

1. Subjects with end-stage renal disease (ESRD) secondary to primary focal segmental glomerulonephritis (FSGS).
2. Inability to comply with study procedures
3. Inability to sign the informed consent
4. Subjects with a significant or active infection
5. Subjects who are pregnant or nursing females
6. Subjects with a history of severe hyperlipidemia not controlled with statins, patients with at total cholesterol of > 400 mg/dl
7. Subjects with a platelet count <100,000mm3 white blood cell (WBC)< 2,000mm3
8. Subjects with severe proteinuria at the time of randomization (>2gm/day)
9. Subjects with more then 2 episodes of acute cellular rejection post transplantation will be excluded from this study
10. An estimated GFR<40 cc/min
11. A history of malignancy during the post-transplant period (other than treated basal cell cancer and/or squamous cell cancer)
12. Subjects, who, due to the existence of a surgical, medical or psychiatric condition, other than the current transplant, which in the opinion of the investigator, precludes enrollment into this trial
13. A history of albumin-creatinine ratio (ACR) during the most recent previous 3 months prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Gallon, MD, Principal Investigator — Northwestern Univesity, Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Stoves J, Lindley EJ, Barnfield MC, Burniston MT, Newstead CG. MDRD equation estimates of glomerular filtration rate in potential living kidney donors and renal transplant recipients with impaired graft function. Nephrol Dial Transplant. 2002 Nov;17(11):2036-7. doi: 10.1093/ndt/17.11.2036. No abstract available. PMID 12401874
- [Background] Gonwa TA, Mai ML, Melton LB, Hays SR, Goldstein RM, Levy MF, Klintmalm GB. End-stage renal disease (ESRD) after orthotopic liver transplantation (OLTX) using calcineurin-based immunotherapy: risk of development and treatment. Transplantation. 2001 Dec 27;72(12):1934-9. doi: 10.1097/00007890-200112270-00012. PMID 11773892
- [Background] Fisher NC, Nightingale PG, Gunson BK, Lipkin GW, Neuberger JM. Chronic renal failure following liver transplantation: a retrospective analysis. Transplantation. 1998 Jul 15;66(1):59-66. doi: 10.1097/00007890-199807150-00010. PMID 9679823
- [Background] Hornberger J, Best J, Geppert J, McClellan M. Risks and costs of end-stage renal disease after heart transplantation. Transplantation. 1998 Dec 27;66(12):1763-70. doi: 10.1097/00007890-199812270-00034. PMID 9884274
- [Background] Goldstein DJ, Zuech N, Sehgal V, Weinberg AD, Drusin R, Cohen D. Cyclosporine-associated end-stage nephropathy after cardiac transplantation: incidence and progression. Transplantation. 1997 Mar 15;63(5):664-8. doi: 10.1097/00007890-199703150-00009. PMID 9075835
- [Background] Myers BD, Ross J, Newton L, Luetscher J, Perlroth M. Cyclosporine-associated chronic nephropathy. N Engl J Med. 1984 Sep 13;311(11):699-705. doi: 10.1056/NEJM198409133111103. PMID 6382005
- [Background] Bennett WM, DeMattos A, Meyer MM, Andoh T, Barry JM. Chronic cyclosporine nephropathy: the Achilles' heel of immunosuppressive therapy. Kidney Int. 1996 Oct;50(4):1089-100. doi: 10.1038/ki.1996.415. No abstract available. PMID 8887265
- [Background] Bennett WM. Insights into chronic cyclosporine nephrotoxicity. Int J Clin Pharmacol Ther. 1996 Nov;34(11):515-9. PMID 8937936
- [Background] Myers BD. Cyclosporine nephrotoxicity. Kidney Int. 1986 Dec;30(6):964-74. doi: 10.1038/ki.1986.280. No abstract available. PMID 3546916
- [Background] Puschett JB, Greenberg A, Holley J, McCauley J. The spectrum of ciclosporin nephrotoxicity. Am J Nephrol. 1990;10(4):296-309. doi: 10.1159/000168123. No abstract available. PMID 2240057
- [Background] Young EW, Ellis CN, Messana JM, Johnson KJ, Leichtman AB, Mihatsch MJ, Hamilton TA, Groisser DS, Fradin MS, Voorhees JJ. A prospective study of renal structure and function in psoriasis patients treated with cyclosporin. Kidney Int. 1994 Oct;46(4):1216-22. doi: 10.1038/ki.1994.387. PMID 7861719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Donor participants were no part of our outcome analysis because their participation was only on the basis of providing blood for testing the immune system of the recipients.
  The analysis of the recipients was intention to treat therefore all recipient participants completed the study period
Period: Overall Study
Arm/Group | Control | Transition to Sirolimus Group
Started | 90 | 185
Completed | 90 | 185
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Donor participants were no part of our outcome analysis because their participation was only on the basis of providing blood for testing the immune system of the recipients.
  The analysis of the recipients was intention to treat therefore all recipient participants completed the study period
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Transition to Sirolimus Group | Total
Number analyzed (Participants) | 90 | 185 | 275
Age, Customized [Mean (Standard Deviation); unit: years]
  Age in years | 39.2 (12.6) | 38.8 (12.5) | 38.9 (12.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex male | 55 | 106 | 161
  Sex female | 35 | 79 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 44 | 83 | 127
  AA | 24 | 37 | 61
  Hispanic | 17 | 45 | 62
  other | 5 | 20 | 25
Region of Enrollment [Number; unit: participants]
  United States | 90 | 185 | 275
HLA mismatch [Mean (Standard Deviation); unit: HLA antigens] — The number of human leukocyte antigens (HLAs) found on the cells of a donor organ but not found on the cells of the organ recipient
  HLA antigens | 3.9 (1.7) | 3.61 (1.82) | 3.8 (1.8)
Donor type [Count of Participants; unit: Participants]
  Living donors | 63 | 130 | 193
  Cadaveric kidneys | 27 | 55 | 82
PRA >20% [Count of Participants; unit: Participants] — A panel-reactive antibody (PRA) is a group of antibodies in a test serum that are reactive against any of several known specific antigens in a panel of test cells or purified HLA antigens from cells. A panel-reactive antibody test (PRA test) is an immunologic test routinely performed by clinical laboratories on the blood of people awaiting organ transplantation.
  This result is the number of participants on the study that had PRA > 20% at the time of Transplantation
  Participants | 14 | 24 | 38
Diabetis mellitus [Count of Participants; unit: Participants] — Number of participants that were diagnosed with Diabetes at the time of Transplantation
  Participants | 26 | 69 | 95
Elevated blood pressure [Count of Participants; unit: Participants] — Number of participant with elevated blood pressure at the time of Transplantation
  Participants | 76 | 158 | 234
Coronary artery disease (CAD) [Count of Participants; unit: Participants] — Coronary artery disease (CAD) occurs when the arteries that supply blood to the heart become hardened and narrowed due to the buildup of cholesterol and other substances, known as plaque
  Participants | 10 | 31 | 41
Smoking [Count of Participants; unit: Participants] | 9 | 29 | 38

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Cellular Rejection
Description: The primary purpose of this research study is to evaluate whether the use of mycophenolate mofetil/Cellcept ® and either tacrolimus/Prograf ® (Group #1) or mycophenolate mofetil/Cellcept ® and sirolimus/Rapamune® (Group #2) impacts the incidence of acute cellular rejection in post-kidney transplant patients. This study will examine whether switching from tacrolimus to sirolimus will better preserve long-term kidney function.
Time Frame: Assessed at 6 Months, 12 Months, 24 Months, months 24 reported
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Transition to Sirolimus Group
Number analyzed (Participants) | 90 | 185
Participants | 7 | 31

2. Secondary Outcome: Renal Allograft Function Calculated With e-GFR and Proteinuria
Description: Evaluate whether CI conversion (tacrolimus→sirolimus) contributes positively or negatively on the renal allograft function calculated with e-GFR and proteinuria
Time Frame: Assessed at 6 Months, 12 Months, 24 Months, months 24 reported
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Control | Transition to Sirolimus Group
Number analyzed (Participants) | 90 | 185
mL/min | 57.6 (20.4) | 58.4 (25.2)

3. Secondary Outcome: Evaluate if CI Conversion Impacts on Lipid Profile, Incidence of Hypertension, Malignancies, and Opportunistic Infections and Post-transplant DM
Description: In addition to monitoring renal allograft function, evaluation will be conducted on the incidence of acute rejection, patient and graft survival, the impact of CI conversion on the lipid profile, the incidence of hypertension, malignancies, opportunistic infections and post-transplant DM (de novo diabetes mellitus).
Time Frame: Assessed at 6 Months, 12 Months, 24 Months, months 24 reported
Measure: Number; unit: number of incidents
Arm/Group | Control | Transition to Sirolimus Group
Number analyzed (Participants) | 90 | 185
number of incidents
  Infections | 33 | 83
  Malignancies | 4 | 9
  Proteinura | 12 | 61
  Hyperlipidemia | 9 | 19
  NODAT | 3 | 2
  BK viremia | 15 | 28
  BK nephropathy | 1 | 5
  Neutropenia | 22 | 35

4. Secondary Outcome: Patient and Graft Survival
Description: This study also reviews the impact of the immunosuppressive medications on patient and graft survival.
Time Frame: Assessed at 6 Months, 12 Months, 24 Months, months 24 reported
Measure: Number; unit: number of incidents
Arm/Group | Control | Transition to Sirolimus Group
Number analyzed (Participants) | 90 | 185
number of incidents
  Kidney transplant loss | 4 | 12
  Patient death | 3 | 10

5. Secondary Outcome: Percentage of Regulatory T Cells
Description: Specifically we reported here the percentage of regulatory T cells that were present in the two groups at 24 months post randomization.
  With peripheral leukocytes taken at baseline (first visit) prior to randomization and at 6, 12 and 24 Months post-randomization, researchers will also review possible modifications of lymphocytes function and of the lymphocytes subpopulations that might have occurred as a consequence of the switch from tacrolimus to sirolimus (randomization).
Time Frame: Assessed at 6 Months, 12 Months, 24 Months, months 24 reported
Measure: Mean (Standard Deviation); unit: % of Treg Cells
Arm/Group | Control | Transition to Sirolimus Group
Number analyzed (Participants) | 90 | 185
% of Treg Cells | 75 (7.1) | 98 (10.8)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Donor participants were no part of our outcome analysis because their participation was only on the basis of providing blood for testing the immune system of the recipients.
  The analysis of the recipients was intention to treat therefore all recipient participants completed the study period
Groups:
- Control: Group 1 will continue immunosuppression medication per standard of care (SOC) at Northwestern by taking mycophenolate mofetil and tacrolimus. Patients were followed for 24 months post randomization
- Transition to Sirolimus: Group 2 will switch immunosuppression medication to taking mycophenolate mofetil and sirolimus. Patients were followed for 24 months post randomization
Arm/Group | Control | Transition to Sirolimus
All-Cause Mortality (participants affected / at risk) | 3/90 | 10/185
Serious Adverse Events (participants affected / at risk) | 42/90 | 117/185
Other Adverse Events (participants affected / at risk) | 58/90 | 135/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=90) | Transition to Sirolimus (N=185)
Renal allograft loss (Renal and urinary disorders) | 4 (4) | 12 (12)
Proteinuria (Renal and urinary disorders) | 12 (12) | 61 (61)
Neutropenia (Blood and lymphatic system disorders) | 22 (22) | 35 (35)
Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=90) | Transition to Sirolimus (N=185)
Infections (Infections and infestations) | 33 (33) | 83 (83)
Hyperlipidemia (Cardiac disorders) | 9 (9) | 19 (19)
Diabetes (Endocrine disorders) | 3 (3) | 2 (3)
BK viremia (Renal and urinary disorders) | 15 (15) | 28 (28)
BK nephropathy (Renal and urinary disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT00866879/Prot_SAP_000.pdf